CLINICAL TRIAL: NCT00947440
Title: An Open-Label, Randomized, Crossover Study to Evaluate the Bioavailability of Two Candidate Tablet Formulations of ABT-072 With Reference to the Capsule Formulation
Brief Title: Evaluation of the Bioavailability of Two ABT-072 Tablet Formulations as Compared to ABT-072 Capsule Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Daniel Cohen, MD/Study Medical Director, Abbott Laboratories
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: M11-056
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-09

CONDITIONS: Hepatitis C
Keywords: Phase 1; Bioavailability
MeSH Terms: conditions — Hepatitis C | interventions — ABT-072

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tablet 1 vs. Capsule (Active Comparator): Single dose of 2 x 50 mg tablets (Tablet 1) vs. 100 mg ABT-072 (contents of capsules) suspended in liquid.
  Interventions: Drug: ABT-072
- Tablet 2 vs. Capsule (Active Comparator): Single dose of 2 x 50 mg tablets (Tablet 2) vs. 100 mg ABT-072 (contents from capsules) suspended in liquid.
  Interventions: Drug: ABT-072

INTERVENTIONS:
Drug: ABT-072 — See arm description for more information

SUMMARY:
The purpose of this study is to assess the bioavailability, safety, tolerability and pharmacokinetics of two tablet formulations as compared to the capsule formulation suspended in liquid.

DETAILED DESCRIPTION:
A single-dose, three period, complete cross-over study to evaluate the relative bioavailability, pharmacokinetics, safety and tolerability of two candidate tablet formulations of ABT-072 when compared to that of the original capsule formulation suspended in liquid as a reference.

ELIGIBILITY:
Inclusion Criteria:

* Overall healthy subjects, non-childbearing females included.

Exclusion Criteria:

* Use of any medications (prescription and over-the-counter), vitamins, or herbal supplements within the 2-week period prior to the first dose of study drug administration or within 10 half-lives of the respective medication, whichever is longer.
* Pregnant or breast-feeding female.
* Positive test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or HIV antibodies (HIV Ab).
* Positive screen for drugs of abuse, alcohol, or cotinine.
* Clinically significant cardiovascular, respiratory (except mild asthma), renal, gastrointestinal, hematologic, neurologic, thyroid, or any uncontrolled medical illness or psychiatric disorder.
* Use of tobacco or nicotine-containing products within the 6-month period preceding study drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the relative bioavailability of two candidate tablet formulations of ABT-072 to that of the capsule formulation. | 4 days post each dose

SECONDARY OUTCOMES:
To evaluate safety and tolerability of two candidate tablet formulations of ABT-072 to that of the capsule formulation. | Through 14 days post last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cohen, MD, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 22384, Waukegan, Illinois, United States